CLINICAL TRIAL: NCT05228197
Title: A Study to Assess the Clinical and Cost-effectiveness of the Galen Prostate Artificial Intelligence Histology System in Diagnosing Clinically Important Prostate Cancer on Prostate Biopsy Tissue.
Brief Title: Imperial Prostate 6 - Cancer Histology Artificial Intelligence Reliability Study.
Acronym: IP6-CHAIROS
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 21CX6823
Record Dates: First submitted 2021-09-24; First posted 2022-02-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; Prostate-Specific Antigen; Artificial Intelligence; Histology
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — H&E stained histology human tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Calibration Stage: Patients referred to hospital urology departments by their GP due to a clinical suspicion of prostate cancer (elevated serum prostate specific antigen [PSA], abnormal feeling prostate on rectal examination). These patients are normally recommended to undergo a prostate MRI as part of standard care.
  Patients will need to meet the Inclusion/Exclusion criteria but in addition, purposive identification of cases with a variety and representative sample of different pathology features are needed for this stage (e.g. normal glands, cancer glands, high-grade PIN, inflammation).
  Interventions: Diagnostic Test: Biopsy & Imaging
- Validation Stage: Patients referred to hospital urology departments by their GP due to a clinical suspicion of prostate cancer (elevated serum prostate specific antigen [PSA], abnormal feeling prostate on rectal examination). These patients are normally recommended to undergo a prostate MRI as part of standard care.
  Patients will need to meet the Inclusion/Exclusion.
  Interventions: Diagnostic Test: Biopsy & Imaging

INTERVENTIONS:
Diagnostic Test: Biopsy & Imaging — H&E stained prostate biopsy slides from standard of care treatment

SUMMARY:
The primary objective is to determine whether the Galen Prostate AI system has sufficient diagnostic accuracy and health economic value to be used for triage of pathology slides within the NHS.

DETAILED DESCRIPTION:
In the UK, about 80-100,000 men every year undergo prostate biopsy to diagnose prostate cancer. This equates to approximately 4 million histology slides; this is estimated to increase to 160,000-200,000 men and up to 6 million slides by 2030 due to rising numbers of men being tested for prostate cancer.

Health Education England and the Royal College of Pathology point to a significant pathology work-force shortage with only 3% of departments having adequate staffing levels and a 10% vacancy rate filled by locums costing £26M every year. By 2021, there will be a 3% decrease of the pathology consultant workforce (40 full-time pathologists); a period of time in which other specialties are expected to see a 13% increase. However, to meet the rising numbers of referrals to pathology departments, it is projected that there will need to be a 3-5% annual growth in the number of pathologists.

Inter-observer variability can occur between pathologists in terms of reporting a diagnosis of clinically important and clinically unimportant prostate cancer by as much as 20% although the differences are smaller when highly expert uro-pathologists are compared. This can lead to inappropriate management of cases.

Galen Prostate AI is a CE-marked deep learning AI-algorithm for prostate needle biopsies that can identify cell types, tissue structures and morphological features for cancer diagnosis. The technology is based on multi-layered convolutional neural networks (CNNs) designed for image classification in which whole-slide imaging is analysed for the detection of tissue areas and then benign versus cancer versus other pathology classification. Compared to almost all competitors, Galen Prostate AI has been tested in ~10 times more tissue samples. Further, Galen Prostate AI is the only algorithm that extends beyond cancer detection/grading to other clinically relevant features (e.g., perineural invasion, high-grade prostatic intraepithelial neoplasia [PIN], inflammation). This AI-algorithm is believed to be the only one in routine clinical deployment - demonstrating technical feasibility and with proven clinical utility.

The proposed study will perform validation in the NHS, for the first time. It is important to stress that this type of algorithm has never been tested on a UK-based population, and in particular, a population that includes a cohort of MRI targeted biopsies, which is now the new diagnostic strategy as it detects clinically relevant prostate cancer in higher percentages than the routine systematic biopsy.

The study is the first and only to address the performance of the AI-based prostate algorithm that extends beyond cancer detection and Gleason grading, by measuring amount of cancer and detecting clinically meaningful features such as perineural invasion in addition to multiple benign structures (e.g. HGPIN, atrophy, inflammation). Given the clinical relevance for such features in the diagnosis process, a study addressing their validation and performance is not only novel, but critical for implementation in routine clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a prostate (either cis-male gender or trans-female gender with no prior hormone use at all).
* Age 18 years or above.
* Undergoing prostate biopsy as a result of an elevated serum PSA or abnormal digital rectal exam, who have undergone a pre-biopsy multi-parametric MRI and advised to undergo prostate biopsies.

(Please note: the Calibration stage requires patients who have already undergone a biopsy and the pathology has been processed over the prior 0 to 12 months).

Exclusion Criteria:

* Unwilling or unable to give consent.
* Any duration or type or dose of androgen deprivation therapy in the 6 months prior to screening.
* Any prior radiotherapy to the prostate or pelvis (including the prostate) or ablation or chemical treatment of the prostate for treating cancer: these types of treatment affect the anatomy of prostate tissue microstructure for which Galen Prostate AI is not currently validated. NB: any treatment for benign enlargement of the prostate is permitted.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Either cis-male gender or trans-female gender with no prior hormone use at all.
Study Population: The target population is patients referred for a prostate biopsy as a result of an elevated serum PSA or abnormal digital rectal exam, who are undergoing or have already undergone prostate biopsies.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Galen Prostate AI | Maximum 6 weeks following enrolment
  Sensitivity, specificity, positive and negative predictive value of Galen Prostate AI on a patient basis for prostate cancer rated Gleason score 7 (ISUP Grade Group >/=2) or greater by consensus pathology review.
Composite Health Outcome (Cost-Consequence Analysis) | Maximum 6 weeks following enrolment
  Includes all the relevant cost and consequences for the Ibex-AI and comparator. Costs: medical equipment, mean cost per diagnosis, primary and secondary care appointments, healthcare professionals' costs, cost of the diagnostic tests and of follow-up testing. Consequences: test accuracy, diagnostic yield, and therapeutic yield.
Composite Health Outcome (Cost-Utility Analysis) | Maximum 6 weeks following enrolment
  Will be presented in the form of an Incremental Cost-Effectiveness Ratio (ICER), a ratio of 'extra cost per extra unit of health outcome' for the intervention vs the comparator.
  Costs: medical equipment, mean cost per diagnosis, primary and secondary care appointments, healthcare professionals' costs, cost of the diagnostic tests and of follow-up testing, implementation costs of adopting the intervention in the NHS, cost of treatment, treatment of adverse effects from the test or treatment, and any monitoring needed before or after the treatment.
  Health outcomes: Quality-adjusted life years (QALY). QALYs will be calculated by estimating the years of life remaining for a patient following diagnosis and weighting each year with a quality-of-life score (EQ-5D questionnaire).

SECONDARY OUTCOMES:
Galen Prostate AI (1) | Maximum 6 weeks following enrolment
  Sensitivity, specificity, positive and negative predictive value of Galen Prostate AI on a slide/biopsy grouping basis (weighted by patient) for prostate cancer rated Gleason score >/=7 (ISUP Grade Group >/=2) by consensus pathology review.
Galen Prostate AI (2) | Maximum 6 weeks following enrolment
  Sensitivity, specificity, positive and negative predictive value of Galen Prostate AI on a patient basis for all prostate cancer.
Galen Prostate AI (3) | Maximum 6 weeks following enrolment
  Area under the receiver operating characteristic curve (AUC) at the patient and slide/biopsy grouping levels for any cancer and clinically significant prostate cancer defined by any Gleason score >/=7 (ISUP Grade Group >/=2).
Galen Prostate AI (4) | Maximum 6 weeks following enrolment
  Agreement of Galen Prostate AI with pathology report for cancer length (mm) on slide/biopsy grouping level and patient level (maximum cancer length).
Galen Prostate AI (5) | Maximum 6 weeks following enrolment
  Agreement of Galen Prostate AI with histology reported percent Gleason Grade pattern 4.
Galen Prostate AI (6) | Maximum 6 weeks following enrolment
  Agreement of Galen Prostate AI with histology reported Gleason score or Grade Group (GG) categories at slide/biopsy grouping level and patient level.
Galen Prostate AI (7) | Maximum 6 weeks following enrolment
  Cancer area (mm2) by slide (Galen Prostate AI only).
Galen Prostate AI (8) | Maximum 6 weeks following enrolment
  Uncalibrated Galen Prostate tool (software) assessed using above primary and secondary metrics.
Pathology Reporting | Maximum 6 weeks following enrolment
  Volume of local pathology reporting (histology slides) on above primary and secondary metrics compared to independent pathology reporting.
Databank Link | Maximum 6 weeks following enrolment
  Databank of scanned high-resolution histology slides and MRI DICOM images linked to clinical parameters for future academic and commercial research into development and validation of diagnostic and prognostic tools for prostate diseases.
Consent to Linkage | Maximum 6 weeks following enrolment
  Number of participants consenting to linkage to national databases for longitudinal healthcare outcomes reporting and correlation to clinical, MR-imaging and histological parameters collected in this study.
Cost-Effectiveness | Maximum 6 weeks following enrolment
  Cost-effectiveness of Galen Prostate system within the NHS (QALYs questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Hashim U Ahmed, Principal Investigator — Imperial College London
Locations (6):
- United Kingdom (6):
  - University Hospitals Coventry and Warwickshire Nhs Trust, Coventry
  - Chelsea and Westminster Hospital Nhs Foundation Trust - Chelsea, London
  - Chelsea and Westminster Hospital Nhs Foundation Trust - West Middlesex, London
  - Imperial College Healthcare Nhs Trust, London
  - University College London Hospitals Nhs Foundation Trust, London
  - University Hospital Southampton Nhs Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No